CLINICAL TRIAL: NCT06464965
Title: A Phase I Clinical Study of Cord Blood-Derived CAR-NK Cells Targeting Claudin18.2 in the Treatment of Advanced Gastric Cancer and Advanced Pancreatic Cancer
Brief Title: Clinical Study of Cord Blood-Derived CAR-NK Cells in Gastric Cancer and Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Zhejiang University (Other); Hangzhou RongGu Biotechnology Limited Company (Unknown)
Responsible Party: Principal Investigator, Liu Yang, MD, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-105
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Pancreas Adenocarcinoma
Keywords: Gastric Cancer; Pancreatic Adenocarcinoma; CAR-NK; Claudin18.2
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CB CAR-NK182 Dose Escalation (Experimental): Participants will receive a lymphodepleting conditioning regimen (FC regimen) followed by three intravenous infusions of Claudin18.2-targeted umbilical cord blood-derived CAR-NK cells (CB CAR-NK182) on days 0, 3, and 7. The study follows a "3+3" dose-escalation design with three planned dose levels.
  Three dose levels: Dose Level 1 (2×10⁶ cells/kg/infusion on days 0, 3, and 7), Dose Level 2 (4×10⁶ cells/kg/infusion on days 0, 3, and 7), Dose Level 3 (8×10⁶ cells/kg/infusion on days 0, 3, and 7). 3-6 subjects will be enrolled per dose level. Each subject will be observed for at least 28 days after the first infusion, with a long-term follow-up period of 2 years post-first infusion.
  Standard "3+3" rules apply for DLT observation and dose escalation decisions.
  Interventions: Biological: CB CAR-NK182; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CB CAR-NK182 — Administered via intravenous infusion on Days 0, 3, and 7.
  Three dose levels are planned:
  Dose Level 1: 2×10^6 cells/kg/infusion Dose Level 2: 4×10^6 cells/kg/infusion Dose Level 3: 8×10^6 cells/kg/infusion
Drug: Cyclophosphamide — Part of the lymphodepletion regimen. Administered at 500 mg/m^2/day on Days -5 to -3 prior to the first CAR-NK cell infusion.
Drug: Fludarabine — Part of the lymphodepletion regimen. Administered at 30 mg/m^2/day on Days -5 to -3 prior to the first CAR-NK cell infusion.

SUMMARY:
Main Objective: To study the maximum tolerated dose (MTD) and dose-dependent toxicity (DLT) of cord blood-derived CAR-NK cells (CB CAR-NK182) targeting Claudin18.2 in patients with advanced gastric cancer and advanced pancreatic cancer.

Secondary Objective: To evaluate the efficacy of CB CAR-NK182 in patients with advanced gastric cancer and advanced pancreatic cancer: overall objective tumor response rate (ORR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS), duration of response (DOR), etc.

To evaluate the CAR-NK amplification and persistence of CB CAR-NK182 in the blood of patients with advanced gastric cancer and advanced pancreatic cancer;

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years (inclusive);
2. Understands and voluntarily signs a written informed consent form, and is willing and able to comply with all trial requirements;
3. Patients with advanced gastric cancer and advanced pancreatic cancer confirmed by histopathology or cytology, who have failed standard treatment or cannot tolerate standard treatment, including but not limited to: pancreatic cancer and gastric cancer;
4. Immunohistochemical (IHC) detection of CLDN18.2, the positive expression of CLDN18.2 in tumors must be ≥ 10%;
5. At least 1 measurable lesion according to RECIST 1.1;
6. ECOG score is 0-1;
7. All toxic reactions caused by previous antineoplastic therapy were resolved to grade 0-1 (according to NCI CTCAE 5.0 edition); Expected survival ≥ 12 weeks;

In addition to the primary disease, no serious hematology, heart and lung, liver and kidney disease, laboratory tests meet the following requirements:

Peripheral blood neutrophil absolute value ≥ 2000/mm3, platelet ≥ 50000/mm3 Serum creatinine ≤ 1.5mg/dL;ALT (alanine aminotransferase)/AST (aspartate aminotransferase) below 2.5 times the upper limit of normal; Total bilirubin ≤ 1.5mg/dL; Cardiac ejection fraction (EF)≥ 50%; International standard ratio (INR) or prothrombin time (PT) below 1.5 times the upper limit of normal; Activated partial coagulation time (aPTT) below 1.5 times the upper limit of normal; 10. Women of childbearing potential must have a negative serum pregnancy test and agree to effective birth control during the treatment phase and within 12 months after injection of CAR-NK cells; Male patients must agree to use effective birth control during the study and for 12 months after injection of CAR-NK cells.

Exclusion Criteria:

1. History of other tumors;
2. Patients who have received CAR-T,CAR-NK,TCR-T and other cell therapy targeting Claudin18.2 within 3 months before study treatment;
3. Patients with hypersensitivity to cell therapy or any related drugs;
4. Active autoimmune diseases;
5. Active infections that cannot be controlled;
6. HIV infection, uncontrolled HBV, HCV and syphilis infections;
7. Have metastatic disease of the central nervous system (CNS), leptomeningeal disease or spinal cord compression;
8. Patients with severe heart disease;
9. Patients with unstable/active ulcers or bleeding from the digestive system;
10. Patients with a history of bleeding or bleeding tendency in the digestive system;
11. Pregnant or lactating women;
12. There are other factors that the researcher believes are not suitable for participating in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
MTD | 1 month
  Maximum Tolerated Dose
DLT | 1 month
  Dose-Dependent Toxicity

SECONDARY OUTCOMES:
ORR | 3 years
  Overall objective tumor response rate
DCR | 3 years
  Disease control rate
PFS | 3 years
  progression-free survival
OS | 3 years
  overall survival
DOR | 3 years
  duration of response

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, M.D., Principal Investigator — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Fanotto V, Cordio S, Pasquini G, Fontanella C, Rimassa L, Leone F, Rosati G, Santini D, Giampieri R, Di Donato S, Tomasello G, Silvestris N, Pietrantonio F, Battaglin F, Avallone A, Scartozzi M, Lutrino ES, Melisi D, Antonuzzo L, Pellegrino A, Torri V, Aprile G. Prognostic factors in 868 advanced gastric cancer patients treated with second-line chemotherapy in the real world. Gastric Cancer. 2017 Sep;20(5):825-833. doi: 10.1007/s10120-016-0681-6. Epub 2016 Dec 27. PMID 28028664
- [Background] Tabernero J, Hoff PM, Shen L, Ohtsu A, Shah MA, Cheng K, Song C, Wu H, Eng-Wong J, Kim K, Kang YK. Pertuzumab plus trastuzumab and chemotherapy for HER2-positive metastatic gastric or gastro-oesophageal junction cancer (JACOB): final analysis of a double-blind, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2018 Oct;19(10):1372-1384. doi: 10.1016/S1470-2045(18)30481-9. Epub 2018 Sep 11. PMID 30217672
- [Background] Thuss-Patience PC, Shah MA, Ohtsu A, Van Cutsem E, Ajani JA, Castro H, Mansoor W, Chung HC, Bodoky G, Shitara K, Phillips GDL, van der Horst T, Harle-Yge ML, Althaus BL, Kang YK. Trastuzumab emtansine versus taxane use for previously treated HER2-positive locally advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma (GATSBY): an international randomised, open-label, adaptive, phase 2/3 study. Lancet Oncol. 2017 May;18(5):640-653. doi: 10.1016/S1470-2045(17)30111-0. Epub 2017 Mar 23. PMID 28343975
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Heinemann V, Ebert MP, Laubender RP, Bevan P, Mala C, Boeck S. Phase II randomised proof-of-concept study of the urokinase inhibitor upamostat (WX-671) in combination with gemcitabine compared with gemcitabine alone in patients with non-resectable, locally advanced pancreatic cancer. Br J Cancer. 2013 Mar 5;108(4):766-70. doi: 10.1038/bjc.2013.62. Epub 2013 Feb 14. PMID 23412098
- [Background] Cappell KM, Kochenderfer JN. Long-term outcomes following CAR T cell therapy: what we know so far. Nat Rev Clin Oncol. 2023 Jun;20(6):359-371. doi: 10.1038/s41571-023-00754-1. Epub 2023 Apr 13. PMID 37055515
- [Background] Khawar MB, Gao G, Rafiq M, Shehzadi A, Afzal A, Abbasi MH, Sheikh N, Afzal N, Ashraf MA, Hamid SE, Shahzaman S, Kawish N, Sun H. Breaking down barriers: The potential of smarter CAR-engineered NK cells against solid tumors. J Cell Biochem. 2023 Aug;124(8):1082-1104. doi: 10.1002/jcb.30460. Epub 2023 Aug 11. PMID 37566723
- [Background] Gowrikumar S, Singh AB, Dhawan P. Role of Claudin Proteins in Regulating Cancer Stem Cells and Chemoresistance-Potential Implication in Disease Prognosis and Therapy. Int J Mol Sci. 2019 Dec 20;21(1):53. doi: 10.3390/ijms21010053. PMID 31861759
- [Background] Kyuno D, Takasawa A, Takasawa K, Ono Y, Aoyama T, Magara K, Nakamori Y, Takemasa I, Osanai M. Claudin-18.2 as a therapeutic target in cancers: cumulative findings from basic research and clinical trials. Tissue Barriers. 2022 Jan 2;10(1):1967080. doi: 10.1080/21688370.2021.1967080. Epub 2021 Sep 5. PMID 34486479